CLINICAL TRIAL: NCT00466583
Title: A Phase 1, Open-Label, Dose Escalation Study Evaluating the Safety and Tolerability of EZN-2968, a Locked Nucleic Acid Antisense Oligonucleotide Against Hypoxia-Inducible Factor-1α, Administered as a Weekly 2-Hour Intravenous Infusion in Adult Patients With Advanced Solid Tumors or Lymphoma
Brief Title: Phase 1 Study of EZN-2968 Weekly in Adult Patients With Advanced Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enzon Pharmaceuticals, Inc. (Industry)
Responsible Party: Noah Berkowitz, MD/Medical Monitor, Enzon Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EZN-2968-01
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-07

CONDITIONS: Carcinoma; Lymphoma
Keywords: Carcinoma, Lymphoma
MeSH Terms: conditions — Carcinoma; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Intravenous EZN-2968 (anti-HIF-1α LNA AS-ODN) — IV infusion of EZN 2968 given in 6 week cycles for (3 weeks on 3 weeks off) until recommended phase 2 dose identified. Up to 3 intensification cohorts will receive the recommended Phase 2 dose of EZN-2968.

SUMMARY:
This is a Phase 1, open-label, non-randomized, dose-escalation study to determine the maximum tolerated dose (MTD), safety, tolerance, and pharmacologic profile of EZN-2968, a locked nucleic acid antisense oligonucleotide against hypoxia-inducible factor 1α administered as a 2-hour intravenous (i.v.) infusion weekly for 3 weeks per 6-week cycle. In patients treated at a recommended Phase 2 dose of EZN-2968, dose intensification will proceed by maintaining the dose, but gradually increasing the number of doses per 6-week cycle. Up to 3 intensification cohorts will receive the recommended Phase 2 dose of EZN-2968.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, non-randomized, dose-escalation study to determine the maximum tolerated dose (MTD), safety, tolerance, and pharmacologic profile of EZN-2968, a locked nucleic acid antisense oligonucleotide against hypoxia-inducible factor 1α (anti-HIF-1α LNA AS ODN) administered as a 2-hour intravenous (i.v.) infusion weekly for 3 weeks per 6-week cycle. In patients treated at a recommended Phase 2 dose of EZN-2968, dose intensification will proceed by maintaining the dose, but gradually increasing the number of doses per 6-week cycle. Up to 3 intensification cohorts will receive the recommended Phase 2 dose of EZN-2968.

ELIGIBILITY:
Inclusion Criteria: Patients must meet all of the following criteria to be eligible for enrollment into the study.

* Histologically or cytologically confirmed diagnosis of advanced and/or metastatic solid tumor or lymphoma (Hodgkin's or non-Hodgkin's)
* Patients who have failed standard therapy and have no known effective therapy available to them
* Patients may have a tumor amenable to biopsy
* Measurable or evaluable disease.
* Age 18 years or older

Exclusion Criteria: Patients meeting any of the following exclusion criteria will not be eligible for enrollment.

* Concurrent serious medical illness
* Known, clinically suspected, or history of central nervous system (CNS) tumor involvement
* Prior chemotherapy, immunotherapy, investigational agent, or other therapy used to treat the cancer within 4 weeks (6 weeks for prior treatment with mitomycin C or nitrosoureas) before the scheduled administration of EZN-2968. Luteinizing hormone-releasing hormone (LHRH) agonist therapy is permitted for patients with hormone refractory prostate cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) of EZN-2968. | January 2011

SECONDARY OUTCOMES:
Determine the pharmacokinetic (PK) profile; Determine the PD profile. | June 2011

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Olszanski, MD, Principal Investigator — Fox Chase Cancer Center; Herbert Hurwitz, MD, Principal Investigator — Duke University; Jose Figueroa, MD, Principal Investigator — Joe Arrington Cancer Center
Locations (3):
- United States (3):
  - Duke University Medical Center, Durham, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas